CLINICAL TRIAL: NCT07090473
Title: Safety of Transcutaneous Electrical Stimulation Potentiating Recovery in Acute Spinal Cord Injury Syndromes
Acronym: STEP-RAISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-40183; CDMRP-SC240091 (Other Grant/Funding Number: US Department of Defense); CDMRP-SC240091P1 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-07-18; First posted 2025-07-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Spinal Cord Injury (SCI); Acute Spinal Cord Injury of Traumatic Origin (tSCI)
Keywords: acute spinal cord injury; transcutaneous spinal cord stimulation; acute rehabilitation; acute traumatic spinal cord injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- active_tSCS (Experimental): active treatment
  Interventions: Device: transcutaneous spinal cord stimulation
- sham_tSCS (Sham Comparator): sham treatment
  Interventions: Device: sham transcutaneous spinal cord stimulation

INTERVENTIONS:
Device: transcutaneous spinal cord stimulation — Transcutaneous spinal stimulation will be delivered using the experimental ARC-EX device (ONWARD Medical), via skin surface electrodes placed over the spine (stimulating electrodes) and bilaterally on the iliac crests (reference electrodes) during the intervention.
  Other Names: non-invasive spinal cord stimulation
  Arms: active_tSCS
Device: sham transcutaneous spinal cord stimulation — For sham transcutaneous spinal stimulation electrodes will be placed on the skin surface over the spine and bilaterally on the iliac crests and will be attached to the experimental ARCEX device (ONWARD Medical), however no electrical current will be delivered.
  Arms: sham_tSCS

SUMMARY:
The goal of this study is to test whether electrical stimulation from the skin surface starting 3 days after spinal cord injury (SCI) is safe and may help patients recover their movement. The main questions it aims to answer are:

* is starting electrical stimulation 3 days post SCI safe?
* can starting electrical stimulation 3 days post SCI help patients recover movement?

This study will be done in two phases. Both phases will be done during the patient's stay in the hospital/intensive care unit (ICU).

In the first phase, participants' will undergo several tests before and after a single treatment. Assessments will be repeated before the patient will go home at around 7 days post injury.

* assessment of the ability to move arms/legs and feel touch or pin prick
* blood and cerebral spinal fluid draws
* assessment of their spinal cord function using electrical stimulation
* receive a single 60-minute continuous electrical stimulation treatment
* patient's safety will be monitored throughout the intervention with the existing standard of care methods in the ICU settings.

In the second phase, researchers will compare active electrical stimulation to sham stimulation to see if active stimulation safely leads to improvement in person's movement ability.

In this second phase, participants' will undergo tests before and after electrical stimulation treatment which will be delivered 5 days in the row. Assessments will be repeated before the patient will go home at around 7 days post injury.

* assessment of the ability to move arms/legs (every day) and feel touch or pin prick (before and after 5 days of treatment)
* blood and cerebral spinal fluid draws (before the first treatment session and before going home)
* assessment of their spinal cord function using electrical stimulation (before the first treatment session and before going home)
* receive daily 60-minute continuous electrical stimulation treatment for 5 days while in ICU
* patient's safety will be monitored throughout the intervention with the existing standard of care methods in the ICU settings.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is often devastating, as many SCI patients are permanently disabled resulting in decades of lost productivity and quality adjusted life years. Patients must largely rely on supportive care, as no Federal Drug Administration (FDA)- approved therapy to treat aSCI exists. Even with early aggressive physical therapy, voluntary movement below the level of the lesion is limited or even absent. There is critical unmet need for strategies to preserve neural function and prevent the host of complications in the hyperacute phase after SCI until discharge to acute rehabilitation.

In the proposed project, Safety of Transcutaneous Electrical stimulation Potentiating Recovery in Acute spinal cord Injury SyndromEs (STEP-RAISE), we will conduct a combined Phase 1 and Phase 2 pilot clinical trial of non-invasive transcutaneous spinal cord stimulation (tSCS), and track the course of neurophysiological recovery following aSCI with granular objective outcome measures to determine whether implementation of early tSCS below the level of lesion can safely augment the functional recovery.

Specific Aims:

Aim 1: Test the safety of tSCS applied below the level of injury to the lumbosacral spinal cord after acute spinal cord injury, starting 72 hours after injury. We hypothesize that there will be no adverse events associated with acute application of tSCS. To assess safety, we will quantify the impacts of tSCS on hemodynamics, spinal cord perfusion pressure (SCPP), and monitor for local skin site reactions.

Aim 2: Demonstrate the proof-of-principle that tSCS application in the acute phase post-injury can potentiate recovery. We hypothesize that tSCS can improve volitional movement and/or sensation acutely after SCI as measured by an improved American Spinal Injury Association Impairment Score (ASIA) score in the presence of tSCS.

Aim 3: Identify novel treatment-related mechanistic biomarkers (exploratory). We hypothesize that there will be fluid-based biomarkers that will change in the setting of tSCS receipt. We will quantify the trajectory of neuronal ubiquitin C-terminal hydrolase L1 (UCH-L1) and glial cell glial fibrillary acidic protein (GFAP) injury markers in the blood and cerebrospinal fluid (CSF) using next generation, high-throughput Olink proteomics (> 5,400 proteins).

Transcutaneous spinal stimulation will be delivered using the experimental ARC-EX device (ONWARD Medical), via skin surface electrodes placed over the spine (stimulating electrodes) and bilaterally on the iliac crests (reference electrodes) during the intervention. The stimulation protocol in this study will be adapted from previously described protocols. Based on previous studies on safety and efficacy of tSCS, we will use biphasic waveforms with a burst frequency of 30 Hz, a carrier frequency of 10 kHz, with a pulse width of 100µs. The neurophysiological assessments described above will be used to characterize the intensity of the stimulation necessary to reach the threshold to elicit muscle responses.

Stimulation will be delivered below the identified motor threshold (subthreshold stimulation intensity) continuously for 60 minutes once a day for 5 days. The intensity of the stimulation will be increased gradually (e.g., 5 mA steps) every session to the motor threshold intensity. Increase in trunk/lower extremity muscle tone will be additionally monitored to assess whether the amplitude of stimulation required to reach motor threshold changes with days post injury + tSCS treatment. If no motor evoked potentials (MEP) can be elicited due to spinal shock, the stimulation intensity will be chosen based on previously reported ranges of effective stimulation, including those observed in our ongoing clinical trial in patients with chronic low back pain (NCT05265000) which provides ranges of maximum tolerable stimulation intensities in individuals without SCI, who have full sensation. The specific stimulation parameters and optimal stimulation intensity will be left to the discretion of the investigators during this experimental treatment. A range of the investigated stimulation parameters will be systematically recorded and will be reported as part of the methodology/study protocol. Participants will be continuously monitored and asked to provide any verbal feedback regarding their sensation of stimulation to ensure there is no pain or discomfort during treatment. For sham stimulation, electrodes will be placed in the same location. The participant will be continually monitored and given similar verbal cues as with the stimulation trials, but no electrical current will be delivered. Participants in both arms will be informed that they may or may not feel the stimulation.

Vital signs will be captured during tSCS and peri-treatment (60 minutes pre- and post-), as well as surface electromyography (EMG).

Exploratory Biomarker Assessments Pre- and Post- treatment Biospecimens for biomarkers will always be drawn after informed consent is signed. We will measure glial fibrillary acidic protein (GFAP) and ubiquitin C-terminal hydrolase L1 (UCH-L1) in blood and CSF on the first day of stimulation prior to the first stimulation session (~72 hours after injury) and on the final day of stimulation (treatment #5) after the last treatment. GFAP and UCH-L1 will be assayed at ZSFG on the Abbott Alinity I Immunoassay system. At those same 2 time points we will also conduct a global discovery proteomic assay on both plasma and CSF. We will use the commercially available high-throughput protein biomarker discovery platform based on Olink's Proximity Extension Assay (PEA), which reliably measures >3,000 proteins using <1mL of biofluid.

Transcutaneous spinal cord stimulation has shown great promise in chronic spinal cord injury rehabilitation medicine through maximizing residual neural circuitry and harnessing neuroplasticity. STEP-RAISE will offer this innovative technology to SCI patients in the acute phase (within days of their injury) to establish the safety, feasibility, and proof-of-concept of this treatment in early recovery. STEP-RAISE offers a creative approach to bringing a rehabilitative intervention to the acute care bedside before the onset of neuro-rehabilitative plateau. This bedside, non-invasive technique has the potential to greatly improve the early management of SCI by offering a bridge to early mobilization which is not currently possible for SCI patients. Given the non-invasive, relatively inexpensive, and portable nature of the technology, tSCS can be deployed in resource limited areas upholding treatment equity for survivors of traumatic SCI.

STEP-RAISE is an essential first step prior to a definitive efficacy trial of tSCS in the ICU. It will provide critical preliminary information that will allow our team to properly design and power such a trial, which if positive, could radically change the paradigm of early rehabilitation in the ICU and change standard of care.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for enrollment in the study of the following criteria apply:

1. Written informed consent is obtained.
2. Acute traumatic cervicothoracic SCI that meets all of the following criteria:

   1. Acute SCI presenting to the hospital within 12 hours of injury
   2. Traumatic non-penetrating SCI
   3. American Impairment Scale (AIS) Grade A, B, or C
   4. International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) neurological level of injury between C4 and T10
3. Aged >/=18 years
4. Admission to Intensive Care Unite (ICU) with lumbar drain in place per standard of care

Exclusion Criteria:

A subject will not be eligible for this study if ANY of the following criteria apply:

1. Subjects classified as AIS D or E
2. Penetrating SCIs or complete transection of the spinal cord
3. Pregnancy
4. Incarceration or police custody
5. Class 2 or Class 3 obesity
6. Any concomitant injury that, in the judgment of the Investigator, interferes with the procedures and examinations required by the study protocol, including but not limited to:

   1. multiple spinal cord lesions
   2. fractures requiring lower extremity casts or splints
   3. skin breakdown or burns over the lumbar spine
   4. profound hemodynamic instability
   5. traumatic brain injury (defined by Glasgow Coma Scale (GCS) <14 at enrollment or inability to participate in exam)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From enrollment to the end of treatment at 7 days post injury
  Number of observed events over the transcutaneous spinal cord stimulation (tSCS) sessions.
  Examples of adverse events (AE) that will be carefully monitored
  * Hemodynamic instability
  * Skin irritation
  * Patient condition deterioration
  * Unanticipated AE
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) motor scores | From enrollment to the end of study at 6 months follow up
  International Standards for Neurological Classification of SCI (ISNCSCI) motor scores; Standardized manual muscle testing is used to assess the strength of each key muscle, typically on a 6-point scale (0-5, 0 - total paralysis to 5 - normal strength with full ROM against gravity and maximal resistance); The motor score is derived by summing the individual muscle grades, with a maximum score of 50 for each upper and lower extremity, and a total maximum score of 100 for both limbs.
  Immediate change in scores with acute tSCS and change in scores from baseline to post treatment and at 6-month follow up will be assessed in the study.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) sensory scores | From enrollment to the end of study at 6 months follow up
  International Standards for Neurological Classification of SCI (ISNCSCI) sensory scores on a 3-point scale to assess sensory function in each dermatome: 0 for absent sensation, 1 for impaired/altered sensation, and 2 for normal sensation. This scoring is done for both light touch and pinprick sensation in each of the 28 dermatomes bilaterally, resulting in a maximum possible score of 112 for each sensation. The sensory level is determined by the most caudal dermatome where sensation is intact for both light touch and pinprick, according to the American Spinal Injury Association.
  Immediate change in scores from baseline vs acute tSCS, post treatment and at 6-months follow up will be assessed.
Motor evoked potentials (MEPs) | From enrollment to post treatment at 7 days post injury
  Single pulse, monophasic spinal cord stimulation will be used to evoke motor potentials. Surface electromyography (EMG) electrodes will be placed on the leg Rectus Femoris (RF), Biceps Femoris (BF), Medial Gastrocnemius (MG) and Tibialis Anterior (TA) muscles, where MEPs will be measured from.
  The data collected will be assessed for MEP presence/elicited (binary measure) and the number of muscles with elicitable MEPs at baseline vs post treatment.
Electromyography (EMG) | From enrollment to study completion at 6 months follow up
  Eight surface electromyography recording electrodes, placed bilaterally over the lower extremity muscles: Rectus Femoris (RF), Biceps Femoris (BF), Medial Gastrocnemius (MG) and Tibialis Anterior (TA) will be used to record motor output (EMG activity) during ISNCSCI assessment.
  Changes in EMG amplitude in the presence of tSCS vs no tSCS (within subject); changes in the number of muscles with EMG output in the presence of tSCS vs no tSCS (within subject) will be analyzed.

SECONDARY OUTCOMES:
Concentration of neuronal (UCH-L1) and glial cell (GFAP) injury markers in blood | From enrollment to the end of treatment at 7 days post SCI
  Blood draw will be collected at baseline post treatment or prior to discharge. Changes in ubiquitin C-terminal hydrolase L1 (UCH-L1) and glial fibrillary acidic protein (GFAP) levels from baseline to post treatment will be assayed on the Abbott Alinity I Immunoassay system. Additionally, plasma will be analyzed using commercially available high-throughput protein biomarker discovery platform based on Olink's Proximity Extension Assay (PEA), which reliably measures >3,000 proteins using <1mL of biofluid
Cerebrospinal fluid (CSF) proteomics | From enrollment to the end of treatment at 7 days post SCI
  CSF will be collected from the lumbar drain tube that is typically placed for acute spinal cord injury management. Changes in protein levels in CSF from baseline to post treatment will be analyzed using commercially available high-throughput protein biomarker discovery platform based on Olink's Proximity Extension Assay (PEA), which reliably measures >3,000 proteins using <1mL of biofluid.
Incidence of neuropathic pain at 6-month follow-up | From enrollment to study completion at 6-months follow up
  DN4 (Neuropathic Pain 4) questionnaire will be used to assess incidence of neuropathic pain at 6-months follow- up in tSCS vs. sham individuals. The DN4 is scored by assigning a value of 1 for each "yes" response and 0 for each "no" response to the 10 questions. A total score is then calculated by summing the scores for all 10 items. A score of 4 or more suggests the presence of neuropathic pain.
Pain Intensity | From enrollment to 6-month follow up
  Pain intensity will be assessed using International Spinal Cord Injury Pain Basic Data Set questionnaire on a 0 - 10 numerical rating scale (ranging from 0 = "No pain" to a maximum of 10 = "Pain as bad as you can imagine").
Quality of Life in Neurological Disorders (Neuro-QoL) scores | At 6-months follow up
  Neuro-QoL questionnaire will be used to assess patients' quality of life. Neuro-QoL questionnaires use a scoring system based on T-scores, where a score of 50 represents the average for a reference population, and a standard deviation is 10 points.
Spinal Cord Independence Measure scores | At 6-month follow up
  Spinal Cord Independence Measure (SCIM) will be administered to assess functional independence. SCIM is a tool used to assess the functional independence of individuals with spinal cord injuries. It focuses on three main areas: self-care, respiration and sphincter management, and mobility. The SCIM score ranges from 0 to 100, with higher scores indicating greater independence.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Saigal, MD, PhD, Principal Investigator — University of California, San Francisco; Anastasia V Keller, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No